CLINICAL TRIAL: NCT00429091
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Dose-Ranging Study of the Safety and Efficacy of ABT-894 in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: A Dose-Ranging Study of the Efficacy of ABT-894 in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Earle Bain, MD, Abbott
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M06-818
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-09

CONDITIONS: Attention-Deficit/Hyperactivity Disorder; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 3-(5,6-dichloropyridin-3-yl)-3,6-diazabicyclo(3.2.0)heptane; Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental)
  Interventions: Drug: ABT-894
- 3 (Active Comparator)
  Interventions: Drug: atomoxetine

INTERVENTIONS:
Drug: ABT-894 — Subjects will take 1 mg QD, 2 mg QD, 4 mg QD, 4 mg BID for up to four weeks.
  Arms: 2
Drug: atomoxetine — Subjects will take 40 mg BID or placebo for up to four weeks.
  Arms: 3
Drug: placebo — Subjects will take BID for up to four weeks
  Arms: 1

SUMMARY:
A Dose-Ranging Study of the Efficacy of ABT-894 in Adults with Attention-Deficit/Hyperactivity Disorder (ADHD)

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for attention-deficit/hyperactivity disorder
* Have voluntarily signed an informed form
* Are between 18 and 60 years of age
* Will use contraceptive methods during the study
* Women must not be pregnant or breast-feeding
* Must be in generally good health
* Are fluent in English

Exclusion Criteria:

* They have a current or past diagnosis of schizoaffective disorder, schizophrenia, obsessive-compulsive disorder, drug-induced psychosis, bipolar disorder, psychotic disorder or mental retardation
* They have a current diagnosis of major depressive episode, generalized anxiety disorder (GAD), or post-traumatic stress disorder (PTSD) or has a clinically significant sleep disorder requiring treatment
* They require ongoing treatment or expected treatment with any psychotropic medication, including anxiolytics, antipsychotics, anticonvulsants, antidepressants, mood stabilizers, nicotine replacement therapies or varenicline
* They require ongoing treatment or expected treatment with Coumadin
* They failed to respond to two or more adequate trials of FDA-approved ADHD medication
* They have taken atomoxetine during the last 3 months
* They have violent, homicidal or suicidal ideation
* They have a significant history of medical diagnoses, seizure disorder, Tourette's syndrome, traumatic brain injury, or a central nervous system (CNS) disease, excluding ADHD
* They have a urine drug screen that is positive for alcohol or drugs of abuse
* They have a history of substance or alcohol disorder during the last 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 243 (Actual)
Dates: Start 2007-01; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
CAARS:Inv Total Score (Sum of Inattentive and Hyperactive/Impulsive Sub-scales) | Final Evaluation of each 4-week Treatment Period

SECONDARY OUTCOMES:
CAARS Inattentive and Hyperactive/Impulsive Sub-scales Scores | Final Evaluation of each 4-week Treatment Period
CAARS ADHD Index | Final Evaluation of each 4-week Treatment Period
CGI-ADHD-S | Final Evaluation of each 4-week Treatment Period
AISRS | Final Evaluation of each 4-week Treatment Period
CAARS:Self | Final Evaluation of each 4-week Treatment Period
TASS | Final Evaluation of each 4-week Treatment Period
FTND | Final Evaluation of each 4-week Treatment Period
QSU-Brief | Final Evaluation of each 4-week Treatment Period
CANTAB cognitive battery | Final Evaluation of each 4-week Treatment Period

CONTACTS AND LOCATIONS:
Overall Officials: Earle Bain, MD, Study Director — Abbott
Locations (22):
- United States (22):
  - Site Reference ID/Investigator# 5965, San Francisco, California
  - Site Reference ID/Investigator# 5955, Wildomar, California
  - Site Reference ID/Investigator# 5974, Orlando, Florida
  - Site Reference ID/Investigator# 5956, West Palm Beach, Florida
  - Site Reference ID/Investigator# 5973, Libertyville, Illinois
  - Site Reference ID/Investigator# 5968, Overland Park, Kansas
  - Site Reference ID/Investigator# 5952, Rockville, Maryland
  - Site Reference ID/Investigator# 5962, Boston, Massachusetts
  - Site Reference ID/Investigator# 5954, Okemos, Michigan
  - Site Reference ID/Investigator# 5970, Troy, Michigan
  - Site Reference ID/Investigator# 5960, Clementon, New Jersey
  - Site Reference ID/Investigator# 5963, Charlotte, North Carolina
  - Site Reference ID/Investigator# 5975, Eugene, Oregon
  - Site Reference ID/Investigator# 5971, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 5957, Charleston, South Carolina
  - Site Reference ID/Investigator# 5972, Austin, Texas
  - Site Reference ID/Investigator# 5959, Bellaire, Texas
  - Site Reference ID/Investigator# 5969, San Antonio, Texas
  - Site Reference ID/Investigator# 5951, Salt Lake City, Utah
  - Site Reference ID/Investigator# 5964, Burlington, Vermont
  - Site Reference ID/Investigator# 5953, Virginia Beach, Virginia
  - Site Reference ID/Investigator# 5958, Bellevue, Washington